CLINICAL TRIAL: NCT00417599
Title: Preventing Overweight in USAF Personnel: Minimal Contact Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, John P. Foreyt, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-10880
Record Dates: First submitted 2006-12-28; First posted 2007-01-01 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Overweight; Obesity
Keywords: Prevention of overweight; Prevention of obesity; Treatment of overweight; Treatment of obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle intervention (Experimental): Behavioral lifestyle intervention versus control group. The Behavioral intervention consists of behavioral lessons delivered over the internet.
  Interventions: Behavioral: Lifestyle Intervention
- control (Experimental): The intervention for the waiting list control group was usual care.
  Interventions: Other: control group

INTERVENTIONS:
Behavioral: Lifestyle Intervention — lifestyle intervention .
  Arms: Lifestyle intervention
Other: control group — waiting list control group
  Arms: control

SUMMARY:
The prevalence of overweight in the United States Air Force (USAF) is about 22%. The objective of this study is to compare the effectiveness of a minimal contact behavioral therapy plus usual care group(MCBT+UC) using a controlled experimental comparison of usual care(UC). Subjects are USAF personnel who are 5lbs below their Maximum Allowable Weight (MAW) and heavier. The primary hypothesis is that: MCBT+UC will have significant weight loss as compared to UC.

DETAILED DESCRIPTION:
The objective of this study is to compare the relative effectiveness of two approaches to weight management, using a controlled comparison experiment. The two approaches are: Minimal Contact Behavior Therapy Plus Usual Care (MCBT+UC) which includes an orientation meeting, provision of a self-help book, use of an interactive weight management web site for 6 months, and 2 brief motivational interviewing telephone follow-ups, plus usual care;and Usual Care (UC) which includes and orientation meeting and usual care (consisting of required USAF annual physical and fitness exam, participation in any mandatory weight loss or fitness programs, and the requirement to stay below a Maximum Allowable Weight [MAW], with penalties or separation as potential contingencies for failure to remain below MAW). The primary outcome is weight loss.Additional outcomes include body mass index, percent body fat, and waist circumference.

ELIGIBILITY:
Inclusion Criteria:

* Within 5 pounds below or equal to their MAW or above MAW according to USAF Weight and height tables
* Access to personal computer with Internet access
* Plan to remain in the local area for one year
* Male or female between the ages 18-55 years

Exclusion Criteria:

* Pregnant, planning to become pregnant or becomes pregnant
* Weight loss of more than 10 pounds in the past 3 months
* No prescription or nonprescription weight-loss medication for at least 6 months prior to screening
* On any medical profile. Specific exclusion includes history of myocardial infarction, stroke, or cancer in the past 5 years, diabetes, angina, and orthopedic or joint problems that would prohibit exercise.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Actual)
Dates: Start 2001-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Body Weight | 1 year

SECONDARY OUTCOMES:
Body Mass Index | 1 year
Percent Body Fat | 1year
Waist Circumference | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: John P Foreyt, Ph.D., Principal Investigator — Baylor College of Medicine
Locations (1):
- Wilford Hall Medical Center AFB, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
See publication: Hunter CM et al Weight management using the internet: a randomized clinical trial. Am J Prev Med 2998;34:119-126

REFERENCES:
- [Derived] Hunter CM, Peterson AL, Alvarez LM, Poston WC, Brundige AR, Haddock CK, Van Brunt DL, Foreyt JP. Weight management using the internet a randomized controlled trial. Am J Prev Med. 2008 Feb;34(2):119-26. doi: 10.1016/j.amepre.2007.09.026. PMID 18201641